CLINICAL TRIAL: NCT01256034
Title: Effects of Preoperative Immunonutrition on Infectious Complication and Th1/Th2 Differentiation in Patients Undergoing Pancreaticoduodenectomy
Brief Title: Effects of Preoperative Immunonutrition in Patients Undergoing Pancreaticoduodenectomy
Acronym: EPIPD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chiba University (Other)
Responsible Party: Principal Investigator, Katsunori Furukawa, MD, PhD, Chiba University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: furukawa2009
Record Dates: First submitted 2010-12-07; First posted 2010-12-08 (Estimated); Results first posted 2012-10-23 (Estimated); Last update posted 2012-10-23 (Estimated); Status verified 2012-09

CONDITIONS: Pancreatic Cancer; Bile Duct Cancer
Keywords: immunonutrition; pancreaticoduodenectomy; Th1; Th2
MeSH Terms: conditions — Pancreatic Neoplasms; Bile Duct Neoplasms | interventions — Long-Term Synaptic Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Active Comparator): preoperative immunonutrition
  Interventions: Dietary Supplement: Oral IMPACT
- Group B (No Intervention): ordinary diet

INTERVENTIONS:
Dietary Supplement: Oral IMPACT — oral supplementation for 5 days (1L/day) before surgery of a formula enriched with arginine, omega-3 fatty acids, and RNA
  Other Names: Oral IMPACT; Ajinomoto Pharma Co., Ltd, Tokyo, Japan
  Arms: Group A

SUMMARY:
The purpose of this study is to determine whether preoperative immunonutrition is effective on infectious complication and Th1/Th2 differentiation in patients with pancreaticoduodenectomy.

DETAILED DESCRIPTION:
The investigators reported that preoperative immunonutrition improve the incidence of postoperative infectious complication in patients after pancreaticoduodenectomy, and modulation of Th1/Th2 differentiation may play important roles in this effect.

Object of this study is to investigate the effects preoperative immunonutrition on incidence of postoperative infectious complication, and Th1/Th2 balance after pancreaticoduodenectomy.

ELIGIBILITY:
Inclusion Criteria:

* patients underwent pancreaticoduodenectomy

Exclusion Criteria:

* age younger than 18 years
* ongoing infection
* gastrointestinal obstruction
* respiratory dysfunction
* cardiac dysfunction
* hepatic dysfunction
* renal failure
* history of recent immunosuppressive or immunological diseases
* preoperative evidence of widespread metastatic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-05; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katsunori Furukawa, MD, Study Director — Chiba University
Locations (1):
- Chiba University, Chiba, Chiba, Japan

REFERENCES:
- [Derived] Aida T, Furukawa K, Suzuki D, Shimizu H, Yoshidome H, Ohtsuka M, Kato A, Yoshitomi H, Miyazaki M. Preoperative immunonutrition decreases postoperative complications by modulating prostaglandin E2 production and T-cell differentiation in patients undergoing pancreatoduodenectomy. Surgery. 2014 Jan;155(1):124-33. doi: 10.1016/j.surg.2013.05.040. Epub 2013 Oct 25. PMID 24589090

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group A | Group B
Started | 25 | 25
Completed | 0 | 0
Not Completed | 25 | 25

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 11 | 20
  >=65 years | 16 | 14 | 30
Age Continuous [Mean (Standard Deviation); unit: years] | 66.4 (7.5) | 65.1 (9.5) | 65.8 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 9 | 14
  Male | 20 | 16 | 36
Region of Enrollment [Number; unit: participants]
  Japan | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Infectious Complication
Time Frame: 30 days
Measure: Number; unit: participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 25 | 25
participants | 7 | 15
Statistical Analysis 1: Comparison: Group A vs Group B; Test type: Superiority or Other; p < 0.05, Chi-squared

2. Secondary Outcome: Plasma IL-6, CRP, Th1/Th2 Balance
Time Frame: 14 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Group A | Group B
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes